CLINICAL TRIAL: NCT02306447
Title: Combined Transcranial and Peripheral Muscle Magnetic Stimulation in Chronic Tinnitus
Acronym: rpms-tinn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., MD, PhD, University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rtms-rpms-tinn
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Tinnitus
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rPMS and rTMS (Experimental): rPMS Stimulation of the neck muscles in five medial-lateral movements starting from the neck: left and right trapezius and deltoid muscle, trapezius and lattissimus dorsi muslce, and over the backbone. 20 stimuli per movement with 2s inter-train interval; four repetitions for each of the five movements; the first 20 trains with a frequency of 5Hz, the second 20 trains at 20Hz; stimulation at individual comfortable level (20-30% stimulator output); round coil.
  rTMS 20Hz stimulation with 2000 stimuli over the left dorso-lateral prefrontal cortex at 110% motor threshold; followed by 1Hz stimulation with 2000 stimuli over the left temporo-parietal cortex; stimulation intensity 110% motor threshold; butterfly coil.
  For stimulation we use MagPro X100 (Medtronic, Denmark).
  Interventions: Device: rPMS and rTMS

INTERVENTIONS:
Device: rPMS and rTMS — rPMS Stimulation of the neck muscles in five medial-lateral movements starting from the neck: left and right trapezius and deltoid muscle, trapezius and lattissimus dorsi muslce, and over the backbone. 20 stimuli per movement with 2s inter-train interval; four repetitions for each of the five movements; the first 20 trains with a frequency of 5Hz, the second 20 trains at 20Hz; stimulation at individual comfortable level (20-30% stimulator output); round coil.
  rTMS 20Hz stimulation with 2000 stimuli over the left dorso-lateral prefrontal cortex at 110% motor threshold; followed by 1Hz stimulation with 2000 stimuli over the left temporo-parietal cortex; stimulation intensity 110% motor threshold; butterfly coil.
  For stimulation we use MagPro X100 (Medtronic, Denmark).

SUMMARY:
Magnetic stimulation of the brain (repetitive transcranial magnetic stimulation) and of neck muscles (repetitive peripheral muscle stimulation) is used to alter tinnitus-related cortical activity and neck muscles tension.

DETAILED DESCRIPTION:
Chronic tinnitus is characterized by several comorbid disorders. One of them is neck and back pain. Here, we investigate the feasibility, safety and clinical efficacy of the combination of repetitive transcranial magnetic stimulation (rTMS) and peripheral muscle stimulation (rPMS) in chronic tinnitus in a pilot study. rTMS is considered to interact with neural tinnitus networks. rPMS is suggested to bring relief to muscle tension. This is an one arm study where explorative analyses will be done with special consideration on patients suffering from neck pain in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bothersome, subjective chronic tinnitus
* Duration of tinnitus more than 6 months

Exclusion Criteria:

* Objective tinnitus
* Treatable cause of the tinnitus
* Involvement in other treatments for tinnitus at the same time
* Clinically relevant psychiatric comorbidity
* Clinically relevant unstable internal or neurological comorbidity
* History of or evidence of significant brain malformation or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorder affecting the brain or prior brain surgery
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse
* Acute neck or back pain
* Neck or back pain of unknown etiology
* Implants in the neck or back, that are sensitive to magnetic fields

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change of tinnitus severity as measured by the tinnitus questionnaire | week 12

SECONDARY OUTCOMES:
Change of tinnitus severity as measured by the tinnitus questionnaire | week 2, week 4, week 12
Change of tinnitus severity as measured by numeric rating scales | week 2, week 4, week 12
Change of depressive symptoms as measured by the major depression inventory | week 2, week 4, week 12
Change in quality of life as measured by the WHOQoL-Bref | week 2, week 4, week 12
Change in neck pain by the neck pain and disability scale | week 2, week 4, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, PhD, Principal Investigator — Department of Psychiatry, University of Regensburg, Germany
Locations (1):
- University of Regensburg, Regensburg, Germany, Germany

REFERENCES:
- [Derived] Vielsmeier V, Schecklmann M, Schlee W, Kreuzer PM, Poeppl TB, Rupprecht R, Langguth B, Lehner A. A Pilot Study of Peripheral Muscle Magnetic Stimulation as Add-on Treatment to Repetitive Transcranial Magnetic Stimulation in Chronic Tinnitus. Front Neurosci. 2018 Feb 20;12:68. doi: 10.3389/fnins.2018.00068. eCollection 2018. PMID 29515350